CLINICAL TRIAL: NCT06323785
Title: Randomised Sham-controlled Trial of Whole-body Hyperthermia for Depression
Brief Title: Whole-body Hyperthermia for Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-D0067
Record Dates: First submitted 2024-02-28; First posted 2024-03-21 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active whole-body hyperthermia (Active Comparator)
  Interventions: Device: Active whole-body hyperthermia
- Sham whole-body hyperthermia (Sham Comparator)
  Interventions: Device: Sham whole-body hyperthermia

INTERVENTIONS:
Device: Active whole-body hyperthermia — Active water-filtered infrared whole-body hyperthermia as described in Janssen et al. (2016)
  Arms: Active whole-body hyperthermia
Device: Sham whole-body hyperthermia — Sham water-filtered infrared whole-body hyperthermia as described in Janssen et al. (2016)
  Arms: Sham whole-body hyperthermia

SUMMARY:
The goal of this clinical trial is to test the efficacy of whole-body hyperthermia in major depression. The main question it aims to answer is:

• Does whole-body hyperthermia alleviate symptoms of depression?

Participants will be randomised to sham or active whole-body hyperthermia. The study will last 6 weeks during which five visits will take place. Depression will be measured repeatedly and biological mechanisms will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* mental capacity to make decisions
* informed consent signed by the subject
* fluent in the German language
* 18-65 years of age
* pre-menopausal women: willing to use birth control or not to engage in sexual intercourse for the duration of the study (the latter only in the case that this corresponds to the habitual lifestyle of this person)
* fulfil DSM-5 criteria for a major depressive episode
* score ≥ 14 on the Hamilton Rating Scale for Depression (HAMD-17; minimum: 0, maximum: 68, higher scores indicate higher depression)
* the major depression is the primary mental disorder

Exclusion Criteria:

* vulnerable subjects
* known or suspected non-compliance, drug or alcohol abuse within the past 2 years
* inability to follow the procedures of the investigation, e.g. due to language problems, psychological disorders, dementia, etc. of the subject
* participation in another investigation with an investigational drug or another MD within the 30 days preceding and during the present investigation
* previous enrolment into the current investigation
* enrolment of the Sponsor-Investigator, her family members, employees and other dependent persons
* contraindications and limitations of the MD as described in the instructions for use
* BMI > 30
* lifetime schizophrenia, lifetime bipolar disorder, current catatonic or psychotic symptoms, current suicidal ideation, current severe claustrophobia, anorexia or bulimia nervosa within the past 5 years
* metallic, silicone, or saline implants
* cardiovascular conditions or problems, including uncontrolled hypertension, congestive heart failure, or documented evidence of coronary artery disease
* chronic conditions/diseases associated with a reduced ability to initiate thermoregulatory cooling, including Parkinson's, multiple sclerosis, central nervous system tumors, and diabetes with neuropathy
* history of peripheral circulatory disease, including peripheral vascular disease and deep vein thrombosis
* history of a cerebral vascular accident
* history of epilepsy or cerebral aneurisms
* cancer in the last five years, except for resected non-melanoma skin cancer
* any clinically significant autoimmune disease
* hemophilia or proneness to bleeding
* fever the day of study intervention
* hypersensitivity to heat
* recent acute joint injury
* enclosed infections, be they dental, in joints, or in any other tissues
* any other medical condition or disorder that is unstable and clinically significant, or that could interfere with the accurate assessment of safety or efficacy of treatment
* intake of medication interfering with thermoregulatory cooling, including barbiturates, diuretics, beta-blockers, and anti-histamines
* intake of psychotropic medication within 2 weeks (8 weeks for fluoxetine)
* need for psychotropic medication during the study period
* current psychotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression (HAMD-17; minimum: 0, maximum: 68, higher scores indicate higher depression) | 1 week
  Depressive symptoms (observer-rated)

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI; minimum: 0, maximum: 63; higher scores indicate higher depression) | 1 week and 6 weeks
  Depressive symptoms (self-reported)
Medical Outcomes Study 36-item short-form health survey (MOS-SF; minimum: 0, maximum: 100, higher scores indicate better health status) | 1 week and 6 weeks
  Quality of life
Hamilton Rating Scale for Depression (HAMD-17; minimum: 0, maximum: 68, higher scores indicate higher depression) | 6 weeks
  Depressive symptoms (observer-rated)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Fischer, PhD, Principal Investigator — University of Zurich
Locations (1):
- University of Zurich, Institute of Psychology, Zurich, Switzerland